CLINICAL TRIAL: NCT02986841
Title: A Phased-Implementation Feasibility and Proof-of-Concept Study to Assess Incorporating the NIDA CTN Common Data Elements (CDEs) Into the Electronic Health Record (EHR) in Large Primary Care Settings ("CDE-EHR-PC" Study), Phase 2
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Massachusetts General Hospital (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 15-01099
Record Dates: First submitted 2016-11-10; First posted 2016-12-08 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a 4-phase study to implement the NIDA (Common Data Elements) Common Data Elements (CDEs) in primary care settings. The study will be conducted at three adult primary care clinics, in two large health systems. Each phase will include deliverables essential to move to the next phase, and an independent Advisory Committee will review progress and make recommendations at each transition about how best to progress to each subsequent phase. Based on progress during earlier phases, the Advisory Committee may recommend expansion to additional clinics or health systems during the second part of Phase 4.

Phase 2 prepares for implementation of the screening and CDS tools as part of routine clinical practice. A key component of this phase is tailoring the screening and CDS tools through an iterative process of usability testing and adaptation of their design. In the KTA framework, this phase corresponds to the 'select, tailor, and implement interventions' step. Simultaneously, investigators will plan for implementation in one clinic of the MSHS system by identifying clinical champions, educating clinic leadership and staff, and conducting a workflow analysis to identify barriers and facilitators of implementation.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adult individuals aged 18 years or older, and employee at a Wave 1 clinic.
* Clinical implementation leaders Clinical implementation leaders are practicing PCPs who provide feedback to the research team and support their colleagues on implementing screening, using the CDS, and carrying out clinical interventions and referrals to address unhealthy substance use. One or two primary care providers will be identified from each clinic site to advise the research team on implementation and to serve as a resource for their colleagues.

Exclusion Criteria:

* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 50 end-user participants will be enrolled. Approximately 5 to 8 end-user participants are required for each cycle of usability testing.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Drug Abuse Screening Test (DAST-10) | 12 Months
  10-item brief screening tool that can be administered by a clinician or self-administered. Each question requires a yes or no response, and the tool can be completed in less than 8 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, MD, MS, Principal Investigator — New York University Medical School
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York